CLINICAL TRIAL: NCT00756353
Title: Out of Care Patient Survey
Brief Title: Survey of Buprenorphine Use Among "Out of Care" Population in France (P04933)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P04933
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Drug Addiction
Keywords: Heroin; Buprenorphine use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Wave 1
- Wave 2

SUMMARY:
This study was a survey of drug users who obtain buprenorphine from the black market and have used buprenorphine during the last month. Subjects were surveyed at various locations (streets, railway stations, etc.) with a few simple questions in order to describe the use of buprenorphine in this "out of care" population.

DETAILED DESCRIPTION:
Participants were found from various places and using a "snow ball" technique.

ELIGIBILITY:
Inclusion Criteria:

* Drug users who have obtained buprenorphine only on the black market or both on black market and in pharmacy.

Exclusion Criteria:

* Patients who have obtained buprenorphine only from the pharmacy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population in this survey includes drug users who are in the "out of care" population, found in various places (streets, railway stations) and via the "snow ball" technique.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The objective of this survey is to describe quantitatively and qualitatively, the use of buprenorphine in the population who obtain buprenorphine only on black market or both on black market and in pharmacy. | Not Applicable, cross-sectional description.

SECONDARY OUTCOMES:
This survey will provide data on patients in regards to their own experience in drug addiction. | Not Applicable, cross-sectional description.